CLINICAL TRIAL: NCT04916301
Title: Developing a Scale for the Psychometric Evaluation of Early Period Mother-Infant Attachment Indicators
Brief Title: Early Period Mother-Infant Attachment Indicators
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Özge Karakaya Suzan, research asistant, Sakarya University
Other Study IDs: developing scale
Record Dates: First submitted 2021-06-01; First posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Early Mother-Baby Attachment
Keywords: Attachment

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Early Mother-Infant Attachment — Early Mother-Infant Attachment Indicators will be observed.

SUMMARY:
The purpose of this study is to develop The Scale for Evaluating Early Mother-Baby Attachment Indicators and to examine its validity and reliability.This is a cross-sectional, methodological, descriptive, and correlational study.The sample of the study for analysis was planned to consist of 130 mothers..The content validity of the scale will assessed by consulting 13 experts in pediatrics, psychiatry and women's health.After the contents of the scale were verified, a pilot test will conducted with a draft scale consisting of 13 items.After the analyzes to be made, it will be tested whether it is a validite and reliable measurement scale.

DETAILED DESCRIPTION:
The behavior of the mother toward her baby in the mother-baby encounter after the birth provides important clues about the bonding process between the mother and the baby in the later period. Therefore, it is important for the nurse responsible for the care of the newborn to carefully observe the mother's behavior to identify the emotional bond between the mother and the baby.Therefore, there is a need for a measurement tool to be developed to be used in the evaluation of early mother-infant attachment, which covers the postnatal period. This scale can enable healthcare professionals to quickly and easily evaluate mother-infant attachment behavior in the early postnatal period. Thus, it can contribute to the early identification of negative attachment behavior that may develop in the future and allow nurses to provide the necessary support. The purpose of this study is to develop The Scale for Evaluating Early Mother-Baby Attachment Indicators and to examine its validity and reliability.

Design and Method Aim This study aims to develop a tool to measure Early Mother-Infant Attachment Indicators and test them psychometrically.

Study Design This is a cross-sectional, methodological, descriptive, and correlational study.

Methodology The development of The Scale for Evaluating Early Mother-Baby Attachment Indicators, the design of the scale, and the phases in its validity are shown in Figure 1. These items include: (1) the preparation and scoping phase; (2) the development of the questionnaire items and rating scale; (3) the content validity; and (4) the pilot study (psychometric evaluation).

Sample/Participants This study will carried out in the XXXX Training and Research Hospital Maternity Service-Infant Team between june and july of 2021. Participants will selected by the random sampling method. The literature states that the number of samples should be at least five times the number of scale items-ideally 10 times the number of items when developing a scale. The number of items in the scale is 13. Accordingly, the study for analysis was planned to consist of 130 mothers. The inclusion criteria were as follows: the participants had to be over 18 years old, had to have volunteered to participate in the study, had to have no health problems related to the newborn, and had to be the mother or the primary care provider.

Data Collection Tools The Sociodemographic Form This form will completed by the mothers while they were in the hospital. It consists of 26 questions about age, the number of children, the maternal educational level, the income levels of the families, and satisfaction with having a baby.

The Scale for Evaluating Early Mother-Baby Attachment Indicators The scale consists of 13 items showing physical and emotional intimacy, exploration, and striving.The content validity of the scale will assessed by consulting 11 experts in pediatrics, psychiatry and women's health.After the contents of the scale were verified, a pilot test will conducted with a draft scale consisting of 13 items Research experts were sent a draft of the Scale for Evaluating Early Mother-Baby Attachment Indicators and a content validity index (CVI) rating form. They were asked to rate the relevance of each item. Relevance was rated on a three-point scale: 1 = not at all relevant, 2 = need to be fixed, 3 = highly relevant. The experts were also encouraged to add comments to each item and to make suggestions for any other item that they deemed necessary but was missing from the instrument. The CVI rating form was created in congruence with best practices for the development of such forms. Rich reviews from experts provided sufficient data for content review. Based on the analysis of the completed CVI forms and the research experts' comments, two scale items were revised.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria were as follows: the participants had to be over 18 years old, had to have volunteered to participate in the study, had to have no health problems related to the newborn, and had to be the mother or the primary care provider.

Exclusion Criteria:

the participants had not to have volunteered to participate in the study, had to have health problems related to the newborn, and had not to be the mother or the primary care provider.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 130 volunteer mothers
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
The Early Mother-Infant Attachment Scale. | one month

CONTACTS AND LOCATIONS:
Overall Officials: Nursan Cinar, Professor, Principal Investigator — Sakarya University

IPD SHARING:
Plan to Share IPD: No